CLINICAL TRIAL: NCT00614809
Title: A Phase II Study of Gefitinib in Benefited Patients With Asymptomatic Brain Metastasis Advanced Non-Small Cell Lung Cancer by Chemotherapy
Brief Title: Efficacy of Gefitinib for Brain Metastasis of Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Yilong,Wu, Guangdong Provincial People's Hospital
Organization: GuangdongPPH (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLC-0703
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer; Brain Metastasis
Keywords: gefitinib; brain metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): non-randomized open-label uncontrolled phase II trial
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib — gefitinib 250mg qd until disease progression or unacceptable toxicity.
  Other Names: IRESSA

SUMMARY:
This is a non-randomized open-label uncontrolled phase II trial evaluating efficacy and toxicity of gefitinib in patients with asymptomatic advanced NSCLC who was benefitted by first line chemotherapy. Patients with stage IV NSCLC who have one or more asymptomatic brain metastasis who was benefitted by first line chemotherapy will receive oral gefitinib 250mg once daily until disease progression or unacceptable toxicity. These patients' direct DNA sequencing of tumor tissue EGFR exons 18-21 will be analyzed The response was evaluated by RECIST criteria after the patient received gefitinib 6 weeks.If the patients present with progress disease of brain metastasis after the therapy of gefitinib, the patients will receive irradiation of brain metastasis.If the response is stable disease,partial response or complete response,he will be examined by brain MRI every 12 weeks.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Histological or cytological documented stage IV NSCLC. Sputum cytology alone is excluded.
2. Extracerebral lesions show stable disease after first line chemotherapy. Patient has recovered from CTCAE grade 3/4 toxicity. Patients who had never received EGFR-TKI or EGFR monoclonal antibody.
3. Patients must be at least 18 years.
4. ECOG Performance Status 0, 1 or 2.
5. Life expectancy of at least 12 weeks.
6. Appraisable disease, the presence of at least three lesions if longest diameter <10 mm by brain MRI.
7. Haemoglobin ³ 10.0 g/dl, Absolute neutrophil count (ANC) ³1.5 x 109/L, platelets ³ 100 x 109/L.
8. Total bilirubin £ 1.5 x upper limit of normal (ULN)
9. ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
10. Creatinine clearance ³ 60ml/min (calculated according to Cockcroft-gault formula).
11. PT-INR/PTT < 1.2 x ULN.
12. Written informed consent.
13. Able to comply with study and follow-up procedures.

Exclusion criteria:

1. Mixed small cell and non-small cell lung cancer histology.
2. Any unresolved toxicity>CTCAE grade 2 from previous anti-cancer therapy.
3. Patients with exposure to biotherapy, immunotherapy within 4 weeks of study entry.
4. Other concurrent anticancer therapy.
5. Patients with exposure to investigational drug therapy outside of this trial.
6. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
7. Any unstable systemic disease (including active infection, hepatic, renal, metabolic disease or seizure disorder requiring medication).
8. Significant cardiovascular event: congestive heart failure >NYHA class 2; unstable angina, active CAD (myocardial infarction more than 1 year prior to study entry is allowed); serious cardiac arrhythmia requiring anti-arrhythmic therapy ( beta blockers or digoxin are permitted) or uncontrolled hypertension.
9. Brain metastases or spinal cord compression, if treated before the start of study treatment, and have any symptoms. Symptoms include signs of increased intracranial pressure ,headache,nausea and vomiting,cognitive or affective disturbances,seizures,and focal neurologic symptoms.
10. History of another malignancy within the last 5 years except cured carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and superficial bladder tumors [Ta, Tis & T1].
11. Pregnant or breast-feeding women.
12. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
13. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

ELIGIBILITY:
Inclusion criteria:

1. Histological or cytological documented stage IV NSCLC. Sputum cytology alone is excluded
2. Extracerebral lesions show stable disease after first line chemotherapy. Patient has recovered from CTCAE grade 3/4 toxicity. Patients who had never received EGFR-TKI or EGFR monoclonal antibody.
3. Patients must be at least 18 years.
4. ECOG Performance Status 0, 1 or 2.
5. Life expectancy of at least 12 weeks.
6. Appraisable disease, the presence of at least three lesions if longest diameter <10 mm by brain MRI.
7. Haemoglobin ³ 10.0 g/dl, Absolute neutrophil count (ANC) ³1.5 x 109/L, platelets ³ 100 x 109/L.
8. Total bilirubin £ 1.5 x upper limit of normal (ULN)
9. ALT and AST < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
10. Creatinine clearance ³ 60ml/min (calculated according to Cockcroft-gault formula).11. PT-INR/PTT < 1.2 x ULN. 12. Written informed consent.13. Able to comply with study and follow-up procedures.

Exclusion criteria:

1. Mixed small cell and non-small cell lung cancer histology.
2. Any unresolved toxicity>CTCAE grade 2 from previous anti-cancer therapy.
3. Patients with exposure to biotherapy, immunotherapy within 4 weeks of study entry.
4. Other concurrent anticancer therapy.
5. Patients with exposure to investigational drug therapy outside of this trial.
6. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
7. Any unstable systemic disease (including active infection, hepatic, renal, metabolic disease or seizure disorder requiring medication).
8. Significant cardiovascular event: congestive heart failure >NYHA class 2; unstable angina, active CAD (myocardial infarction more than 1 year prior to study entry is allowed); serious cardiac arrhythmia requiring anti-arrhythmic therapy ( beta blockers or digoxin are permitted) or uncontrolled hypertension.
9. Brain metastases or spinal cord compression, if treated before the start of study treatment, and have any symptoms. Symptoms include signs of increased intracranial pressure ,headache,nausea and vomiting,cognitive or affective disturbances,seizures,and focal neurologic symptoms.
10. History of another malignancy within the last 5 years except cured carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and superficial bladder tumors [Ta, Tis & T1].
11. Pregnant or breast-feeding women.
12. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
13. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Time of asymptomatic brain metastasis turn into symptomatic brain metastasis | 12/2007~12/2010

SECONDARY OUTCOMES:
To determine objective response (CR+PR), time to progression, 6-month survival and 1-year survival,safety. | 12/2007~12/2010

CONTACTS AND LOCATIONS:
Overall Officials: Wu yilong, MD, Principal Investigator — Director of cancer center of Guangdong PPH